CLINICAL TRIAL: NCT00160914
Title: Childhood Obesity: Variations in Management
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Collaborators: The Nathan Cummings Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11408B
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
Keywords: Childhood obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Identification/management of childhood obesity (behavior) — In this project, we plan to conduct a national survey of pediatricians to assess common strategies for identification and management of childhood obesity, along with pediatricians' attitudes and beliefs about childhood obesity.

SUMMARY:
Childhood obesity has been described as a growing national epidemic. Between 1980 and 1994 the prevalence of childhood obesity doubled with 10% to 15% of children and adolescents being obese. Childhood obesity has both immediate and long-term detrimental consequences for health and well-being. Obese children are at increased risk for coronary heart disease, type 2 diabetes, and hypertension. Obese children are more likely to be at risk for psychological stress and disturbed body image. Moreover, obese children are more likely to become obese adults, especially if weight reduction has not occurred by the end of adolescence.

The pediatrician is in an ideal position to assess and manage childhood obesity. Recently, guidelines have been established for the assessment and treatment of childhood obesity. These "best practice" guidelines include recommended diagnostic criteria, assessment of contributing factors such as diet and lifestyle, family history, and treatment choices. Although these guidelines have been introduced little is known about pediatricians' actual practice patterns and their beliefs concerning childhood obesity.

Project Description I plan to conduct a national survey of pediatricians to assess common strategies for the identification and management of childhood obesity, along with pediatricians' attitudes and beliefs about childhood obesity. In consultation with a panel of practicing general pediatricians and survey research experts, I plan to develop a survey that measures pediatricians' beliefs about the causes and consequences of childhood obesity, its prevalence in their practice settings, their approaches to diagnosis and management, and resources available for treatment. The survey will be administered to a randomly selected national sample of approximately 600 practicing general pediatricians. The response rate is expected to be approximately 60% or 360 pediatricians. The survey results will help to assess the degree to which recommended practice guidelines are being implemented, identify pediatricians' beliefs and attitudes that might serve as barriers to optimal care, and suggest areas for continuing medical education. The proposed time frame for the study is two years.

DETAILED DESCRIPTION:
Project Goals

Year One

* Develop and Pilot Test Survey. The Pediatrician Survey will be designed to assess both practice patterns and attitudes/beliefs pertaining to childhood and adolescent obesity. From a review of the literature and the recently published guidelines, along with interviews with practicing pediatricians, we will generate items that assess relevant diagnostic and therapeutic approaches to childhood obesity, including patient and physician demographic data. We will also thoroughly review the literature to identify attitudes and beliefs that may impact pediatricians approaches to obesity management. The survey will be pilot tested with a small sample of practicing pediatricians, and appropriate modifications in the survey will be made.
* Select Sample. We will use the American Academy of Pediatrics Fellowship Directory to identify a national pool of practicing pediatricians. To allow us to assess any regional differences in practice patterns, we will stratify the pool of practicing pediatricians by geographic region and randomly select 150 pediatricians from within each of four geographic regions. This will allow us to survey a total of 600 practicing pediatricians.
* Mail Surveys. Using addresses provided by the Directory, we will send surveys via mail to selected pediatricians. All mailings will be coded and entered into a computerized master list that will facilitate tracking of surveys received and follow-up. Surveys sent and received will be tracked. Based on prior research experience, we expect an initial response rate of approximately 50%. One month after the initial mailing, we will conduct a second mailing to non--responders, sending a reminder postcard requesting the completion and return of the survey. Two months after the initial mailing, a second letter and survey will be sent to those who still have not responded. With this method, we expect a final response rate of 60%

Year Two

• Data Entry and Analysis. Data from returned surveys, including respondent demographic characteristics, practice structure and setting, practice patterns, and attitudes/beliefs will be entered into a database for subsequent analysis. Data will be double-entered and checked for accuracy. Data analysis will consist of establishing psychometric properties of attitude and belief measures, examining frequencies of responses to, individual items, looking for trends across geographic regions, and assessing common approaches to the diagnosis and management of childhood obesity. Moreover, we will analyze the data to determine the relationship of attitudes/beliefs and practice patterns. We anticipate that we will identify a number of important variations in the diagnosis and management of childhood obesity. We also expect to identify a number of personal and systems-related barriers to treatment of childhood obesity. For example, we expect that pediatricians with more recent training will have more optimistic attitudes toward successful management of childhood obesity. We also expect to find variations in reimbursement and clinic resources, and that these will impact pediatricians' approaches.

ELIGIBILITY:
Inclusion Criteria:

* Practicing general pediatricians

Exclusion Criteria:

* Non practicing general pediatricians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Practicing general pediatricians
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2001-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janis Mendelsohn, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Flegal KM, Carroll MD, Kuczmarski RJ, Johnson CL. Overweight and obesity in the United States: prevalence and trends, 1960-1994. Int J Obes Relat Metab Disord. 1998 Jan;22(1):39-47. doi: 10.1038/sj.ijo.0800541. PMID 9481598
- [Background] Lauer RM, Connor WE, Leaverton PE, Reiter MA, Clarke WR. Coronary heart disease risk factors in school children: the Muscatine study. J Pediatr. 1975 May;86(5):697-706. doi: 10.1016/s0022-3476(75)80353-2. PMID 1133650
- [Background] Drash A. Relationship between diabetes mellitus and obesity in the child. Metabolism. 1973 Feb;22(2):337-44. doi: 10.1016/0026-0495(73)90185-6. No abstract available. PMID 4687958
- [Background] Londe S, Bourgoignie JJ, Robson AM, Goldring D. Hypertension in apparently normal children. J Pediatr. 1971 Apr;78(4):569-77. doi: 10.1016/s0022-3476(71)80457-2. No abstract available. PMID 5555589
- [Background] French SA, Story M, Perry CL. Self-esteem and obesity in children and adolescents: a literature review. Obes Res. 1995 Sep;3(5):479-90. doi: 10.1002/j.1550-8528.1995.tb00179.x. PMID 8521169
- [Background] Serdula MK, Ivery D, Coates RJ, Freedman DS, Williamson DF, Byers T. Do obese children become obese adults? A review of the literature. Prev Med. 1993 Mar;22(2):167-77. doi: 10.1006/pmed.1993.1014. PMID 8483856
- [Background] Barlow SE, Dietz WH. Obesity evaluation and treatment: Expert Committee recommendations. The Maternal and Child Health Bureau, Health Resources and Services Administration and the Department of Health and Human Services. Pediatrics. 1998 Sep;102(3):E29. doi: 10.1542/peds.102.3.e29. PMID 9724677
- [Background] American Academy of Pediatrics. Fellowship Directory. Elk Grove Village, IL: American Academy of Pediatrics., 2001.
- [Background] Dietz WH, Nelson A. Barriers to the treatment of childhood obesity: a call to action. J Pediatr. 1999 May;134(5):535-6. doi: 10.1016/s0022-3476(99)70235-0. No abstract available. PMID 10228284